CLINICAL TRIAL: NCT00742534
Title: Phase 1 Intravenous Citrulline for the Prevention of Bronchopulmonary Dysplasia in Preterm Infants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never began
Sponsor: Vanderbilt University (Other)
Responsible Party: Frederick E. Barr, MD, MSCI, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPD2008
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Prematurity; Lung Disease; preterm infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intravenous L-Citrulline — This is a classic dose escalation using initial doses of 10 mg/kg of intravenous citrulline and advancing the dose by 10 mg/kg every 3 patients for a target peak plasma citrulline concentration of 100 umol/L. This regimen will be adjusted with pharmacokinetic data as it becomes available so that it may be adjusted to maintain appropriate serum levels of the urea cycle precursors and NO metabolites of interest.

SUMMARY:
Premature infants are at risk for developing bronchopulmonary dysplasia (BPD). L-citrulline may decrease that risk, but we do not know the safety or dose of this drug for use in premature babies. The purpose of this study is to determine the safety and optimal dose of intravenous L-citrulline in premature infants.

DETAILED DESCRIPTION:
This is a prospective phase I study of the safety, pharmacokinetics, and optimal dose of intravenously administered L-citrulline in premature infants born at 24 to 29 weeks estimated gestational age (EGA) and who are at risk for bronchopulmonary dysplasia (BPD). This is a classic dose escalation using initial doses of 10 mg/kg of intravenous citrulline and advancing the dose by 10 mg/kg every 3 patients for a target peak plasma citrulline concentration of 100 umol/L. These infants will undergo intense hemodynamic monitoring and have intermittent blood sampling to determine levels of amino acids and nitric oxide metabolites. From this, we will determine citrulline pharmacokinetics including half life, clearance, and volume of distribution. Intravenous L-citrulline will be provided by Asklepion Pharmaceuticals and mixed by the Investigational Drug Service of the Vanderbilt Hospital Clinical Pharmacy. The study will be monitored closely by a data safety monitoring board (DSMB) consisting of clinicians not involved with this study.

ELIGIBILITY:
Inclusion Criteria:

* 24-29 Weeks Gestation
* Respiratory Distress requiring intubation and mechanical ventilation or positive pressure oxygen at 24 hours of life
* Parents willing and able to sign consent

Exclusion Criteria:

* Congenital malformation
* Suspected genetic or metabolic syndrome
* Surgical condition
* Life expectancy < 24 hours
* Pre-existing, sustained hypotension
* Birth weight < 500 grams
* Any condition which, in the opinion of the investigator, will interfere with the study objectives.

Ages: 2 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics and dose finding in preterm infants with BPD | Surrounding Dose

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E Barr, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States